CLINICAL TRIAL: NCT01938313
Title: Comparison of ERAS (Early Recovery After Surgery) Protocol With Conventional Protocol After Laparoscopic Gastrectomy: A Prospective Randomized Controlled Trial (Phase II Study))
Brief Title: Early Recovery After Surgery (ERAS) Versus Conventional Protocol After Laparoscopic Gastrectomy
Acronym: ERAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-ERAS-GC-PII
Record Dates: First submitted 2012-07-15; First posted 2013-09-10 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; ERAS (early recovery after surgery); fast track; laparoscopic gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERAS perioperative cares (Active Comparator): Patients planned to undergoing laparoscopic gastrectomy, following the ERAS protocols.
  Interventions: Procedure: ERAS perioperative cares
- Conventional perioperative cares (Active Comparator): Patents will be managed by our hospital's critical pathways.
  Interventions: Procedure: Conventional perioperative cares

INTERVENTIONS:
Procedure: ERAS perioperative cares — 1. Patient's preoperative counseling & education before surgery
  2. No Bowel preparation
  3. Oral Carbohydrate Solution (OCS) loading until 2hours before surgery
  4. Fluid restriction & Management by pulse contour analysis or transesophageal doppler
  5. Early mobilization
  6. Early oral feeding (postoperative 1 day - sips of water, 2 days - semifluid diet (SFD), 3 days - soft blended diet (SBD))
  7. Epidural patient controlled analgesics (no opioids analgesics)
  8. Postoperative Nausea Active Control
  9. Thromboembolism prophylaxis by low molecular weighted heparin (LMWH)
  10. Perioperative High content Oxygen therapy
  11. No drain insertion
  12. No Levin tube
  13. Patients will be discharged at POD#4 if there's no problem.
  Arms: ERAS perioperative cares
Procedure: Conventional perioperative cares — 1. No Patient's preoperative counseling & education before surgery
  2. Bowel preparation
  3. No Oral Carbohydrate Solution (OCS) loading until 2hours before surgery
  4. Conventional Fluid Management by clinical signs (Urine output, heart rate etc.)
  5. Conventional Mobilization
  6. Conventional oral feeding (POD#2 SOW, #3 SFD, #4 SBD)
  7. IV PCA
  8. Postoperative Nausea Control if needed
  9. No Thromboembolism prophylaxis
  10. No or Low Content Oxygen therapy
  11. Routine drain insertion
  12. Levin tube insertion if needed
  Arms: Conventional perioperative cares

SUMMARY:
Enhanced Recovery After Surgery (ERAS) programs have been introduced with purposes of reducing the surgical stress response and obtaining optimal recovery after surgery.

DETAILED DESCRIPTION:
There is strong evidence of the usefulness of the ERAS programs in patients undergoing colorectal surgery in terms of significantly reduced postoperative complications and shorter length of hospital stay, compared to the patients of conventional treatment.

However, few studies exist about the implication of ERAS programs in the laparoscopic gastrectomy.

The aim of this study was to compare the recovery rate, morbidity, and quality of life in the patients undergoing laparoscopic gastrectomy for gastric cancer, receiving either ERAS protocol or conventional postoperative cares.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American Society of Anesthesiologists (ASA) scores < 3
* 20 < Age < 80
* Gastric cancer, adenocarcinoma, possible to perform laparoscopic distal gastrectomy
* Informed consent
* No other treatment (Radiation, Chemotherapy or Immunotherapy) on this gastric cancer or other type of cancer.
* No systemic inflammatory disease

Exclusion Criteria:

* Emergency operation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recovering Rate | 4 days after surgery
  1. Tolerance of diet for 24 hours A. Able to eat one third of more of soft-blend meal without abdominal discomfort, bloating, nausea, or vomiting
  2. Analgesic-free (oral or IV analgesic drugs not necessary after cessation of PCA)
  3. Safe ambulation (ambulation of 600m without assistance)
  4. Afebrile status without major complications (fever defined as body temperature greater than 37.5)
     * Above total 4 criteria should be satisfied for the evaluation of complete recovery.

SECONDARY OUTCOMES:
Postoperative length of hospital stay | up to 4 weeks after surgery
Time to tolerance of a full diet | up to 1 month after surgery
Time to first bowel motion Time to first bowel motion | up to 7 days after surgery
Complications during the admissionTime to first bowel motion | up to 30 days after surgery
Readmission rate | up to 30 days after surgery
Pain scores based on a visual analog scale the day of surgery and the subsequent 3 days | up to 3 days after surgery
  postoperative 2hours, 6 hours, 1 days, 2 days, 3 days
Quality of life | up to 1 month after surgery
  European organization for research and treatment of cancer (EORTC) and gastrointestinal quality of life index (GIQLI) questionnaire on postoperative 5 days, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Ho Kim, M.D., Ph.D., Principal Investigator — Department of Surgery, SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Geynggi, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang SH, Lee Y, Min SH, Park YS, Ahn SH, Park DJ, Kim HH. Multimodal Enhanced Recovery After Surgery (ERAS) Program is the Optimal Perioperative Care in Patients Undergoing Totally Laparoscopic Distal Gastrectomy for Gastric Cancer: A Prospective, Randomized, Clinical Trial. Ann Surg Oncol. 2018 Oct;25(11):3231-3238. doi: 10.1245/s10434-018-6625-0. Epub 2018 Jul 26. PMID 30051365